CLINICAL TRIAL: NCT03474432
Title: SOLEMN Study - Synergy Optical Coherence Tomography in Left Main PCI
Acronym: SOLEMN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of enrollment.
Sponsor: Jesse Brown VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mladen I. Vidovich, Associate Professor of Medicine, University of Illinois at Chicago and Chief of Cardiology, Jesse Brown VA Medical Center, Jesse Brown VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JBVA-MIV-001
Record Dates: First submitted 2018-03-02; First posted 2018-03-22 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Percutaneous Coronary Intervention; Optical Coherence Tomography; In-stent Coronary Artery Restenosis
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Optical Coherence Tomography (Other): Patients who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure will be approached for the study and enrolled if eligible.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — OCT will be performed with the St. Jude OCT system. Detection of metallic stent struts will be performed automatically with manual adjustments made as necessary. Stent area tracings will be automatically performed by interpolated contours connecting the center point of the luminal surface of each detected metallic strut. Stent expansion will be determined as the minimum stent area divided by the average reference lumen area and presented as a percentage. Neo-intimal hyperplasia (NIH) area will be determined in follow-up examinations as the area between the stent and lumen contours. Incomplete stent apposition (ISA) area will be determined as the area between the stent contour and the lumen contour at the site of malapposed struts, in a region not overlying a side branch ostium.
  Other Names: Dragonfly OPTIS Imaging Catheter

SUMMARY:
BACKGROUD:

Percutaneous coronary intervention (PCI) is increasingly used to treat unprotected left main coronary artery stenosis. Protected LM PCI is considered standard of care in most centers.

OCT allows for precise determination of stent placement, stent expansion and apposition. The pattern of vessel healing can be very precisely studied if immediate post-stent implantation OCT/IVUS data is compared to the 6-month post-PCI interval.

While OCT cannot be optimally used for ostial lesion imaging, IVUS can be used to image ostial lesions/stent placement.

Optimal and consistent vessel healing is particularly important in LM PCI where stent thrombosis is a potential complication with serious adverse outcome.

HYPOTHESIS:

Due to the absorption of the polymer of the Boston Scientific Synergy Stent over time, early strut coverage patterns and timeline may be different than previously observed in DES and BMS stents in LM PCI. Late acquired stent malapposition (LASM) is expected to differ from previous observations with traditional DES/BMS.

Stent coverage in LM PCI will be studied with OCT or IVUS at six and 12 months and compared to OCT or IVUS at the time of stent implantation.

OCT/IVUS data will be analyzed in a core lab (CRF) and correlated with clinical outcomes at 6 and 12 months.

DETAILED DESCRIPTION:
The proposed study is a multicenter, observational, prospective, single-arm study of stent strut coverage of patients undergoing LM PCI.

Baseline quantitative coronary analysis (QCA) will be performed at the time of stent implantation.

Stent coverage in LM PCI will be studied with OCT at 3 and 12 months and compared to baseline OCT at the time of stent implantation.(31, 32)

OCT/data will be analyzed in a core lab (CTC CRF) and correlated with clinical outcomes at 3 and 12 months.

Primary Endpoint

• 3-month stent strut coverage in LM PCI

Secondary Endpoints

* 12-month stent strut coverage in LM PCI
* 3-month late acquired stent malapposition (LASM)
* 12-month late acquired stent malapposition (LASM)
* One-month LM Synergy stent safety
* 1-, 3- and 12-month MACE
* 1-, 3- and 12-month Stent Thrombosis (ST) (ARC definition)

  75 patients undergoing LM PCI (protected or unprotected) with Boston Scientific Synergy™ stent.

The goal is to enroll 75 patients from up to 10 VA sites and an enrollment period of 3 years, each site is expected to include 7-10 patients during the study period.

After a total of 75 patients are enrolled the study will be closed for further enrollment.

Eligible patients will be screened at each participating center and those who had undergone LM PCI with Boston Scientific Synergy™ stent and where OCT was performed during the index procedure will be eligible. The index procedure may be performed by any interventional cardiologist - this is specifically needed in order to maintain equipoise on the part of stent choice and use of OCT.

At the end of the study enrollment period, the proportion of patients at each site treated with Synergy stents vs. non-Synergy stents and the proportion of patients that underwent OCT imaging during LM PCI will be collected.

Eligible patients will be approached and consented for inclusion in the SOLEMN trial after the initial procedure.

Study Duration

Patients will be followed for 12 months after the index procedure. At one month, clinical follow-up will be performed (clinic or telephone). At 3 months, the angiography and OCT will be performed. At 12 months, the final angiography and OCT will be performed. No further follow-up is planned after completion of the 3- and 12-month angiography and OCT.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or greater;
* Left Main CAD, defined as ≥ 50% diameter stenosis and amenable to re-vascularization by PCI;
* Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
* Ability to comply with minimum of 6 months of DAPT after the index procedure.
* Unprotected Left Main PCI
* Protected Left Main PCI

Exclusion criteria:

* Coexisting conditions that limit life expectancy to less than 12 months or that could affect patient's compliance with the protocol;
* Serum creatinine greater than 2.0 mg/dL;
* Cardiogenic shock;
* STEMI;
* Non-STEMI, if the cardiac troponin is not stable or starting to decline;
* Pregnancy;
* Inability to take dual antiplatelet therapy for 6 months;
* Any target lesion with previously placed stent.
* Patients disqualified for CABG surgery.
* Contraindications for OCT use:

  1. Bacteremia or sepsis
  2. Major coagulation system abnormalities
  3. Severe hemodynamic instability or shock
  4. Patients diagnosed with coronary artery spasm
  5. Acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mladen I Vidovich, MD, Principal Investigator — Jesse Brown VA Medical Center
Locations (13):
- United States (13):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - VA Long Beach Healthcare, Long Beach, California
  - San Francisco VA, San Francisco, California
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Jesse Brown VAMC, Chicago, Illinois
  - VA Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Oklahoma City VA Health Care System, Oklahoma City, Oklahoma
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - San Antonio VA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Optical Coherence Tomography: Patients who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure will be approached for the study and enrolled if eligible.
  Optical Coherence Tomography: OCT will be performed with the St. Jude OCT system.
  Detection of metallic stent struts will be performed automatically with manual adjustments made as necessary. Stent area tracings will be automatically performed by interpolated contours connecting the center point of the luminal surface of each detected metallic strut. Stent expansion will be determined as the minimum stent area divided by the average reference lumen area and presented as a percentage. Neo-intimal hyperplasia (NIH) area will be determined in follow-up examinations as the area between the stent and lumen contours. Incomplete stent apposition (ISA) area will be determined as the area between the stent contour and the lumen contour at the site of malapposed struts, in a region not overlying a side branch ostium.
Period: Overall Study
Arm/Group | Optical Coherence Tomography
Started | 12
Completed | 6
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Left Main Coronary Artery stenosis
Arm/Group | Optical Coherence Tomography
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: The Stents Analyzed for Strut Coverage in LM Percutaneous Coronary Intervention (PCI)
Description: The stents from 6 participants were analyzed for strut coverage, which is specifically defined as Percentage of Uncovered Stent Struts. The Percentage of Uncovered Stent Struts is the number of struts without distinct overlying tissue, in which the luminal reflection of the strut surface is directly interfacing with the lumen, divided by total number of analyzable struts.
Time Frame: 3 Months
Population: 6 participants had stents analyzed at 3 months.
Measure: Median (Inter-Quartile Range); unit: Percentage of Uncovered Stent Struts
Units Other Than Participants: Stents
Arm/Group | Optical Coherence Tomography
Number analyzed (Participants) | 6
Number analyzed (Stents) | 6
Percentage of Uncovered Stent Struts | 93.8 [86.3 to 95.0]

2. Secondary Outcome: The Stents Analyzed for Strut Coverage in LM Percutaneous Coronary Intervention (PCI)
Description: The stents from 2 participants were analyzed for strut coverage, which is specifically defined as Percentage of Uncovered Stent Struts. The Percentage of Uncovered Stent Struts is the number of struts without distinct overlying tissue, in which the luminal reflection of the strut surface is directly interfacing with the lumen, divided by total number of analyzable struts.
Time Frame: 12 month
Population: 2 participants had data analyzed at 12 months.
Measure: Median (Inter-Quartile Range); unit: Percentage of Uncovered Stent Struts
Units Other Than Participants: Stents
Groups:
- Optical Coherence Tomography: Patients who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure will be approached for the study and enrolled if eligible.
  Optical Coherence Tomography: OCT will be performed with the St. Jude OCT system.
  Detection of metallic stent struts will be performed automatically with manual adjustments made as necessary. Stent area tracings will be automatically performed by interpolated contours connecting the center point of the luminal surface of each detected metallic strut. Stent expansion will be determined as the minimum stent area divided by the average reference lumen area and presented as a percentage. Neo-intimal hyperplasia (NIH) area will be determined in follow-up examinations as the area between the stent and lumen contours. Incomplete stent apposition (ISA) area will be determined as the area between the stent contour and the lumen contour at the site of malapposed struts, in a region not overlying a side branch ostium.
  Between July 11, 2018 and December 31, 2019, 12 participants with 13 treated lesions were enrolled. Two patients were lost to follow-up, two patients withdrew consent due to living too remotely to follow up, one patient's imaging data was unreadable upon analysis, and one patient was withdrawn by an investigator prior to follow-up for worsening renal function. Six participants with 7 treated lesions had at least 3-month follow-up data and 2 patients had 12-month data available.
Arm/Group | Optical Coherence Tomography
Number analyzed (Participants) | 2
Number analyzed (Stents) | 2
Percentage of Uncovered Stent Struts | 94.7 [93.6 to 95.7]

3. Secondary Outcome: 3-month Persistent Stent Malapposition
Description: Malapposition is determined by measuring of the distance from the center of blooming to the nearby endoluminal surface of the intima. Malapposition is defined as a measured distance than the total thickness of the stent metal plus polymer of the stent (greater than 200 µm). Malapposition was considered persistent, since was already present at baseline.
Time Frame: 3 month
Population: Number of participants with persistent stent malapposition at 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Optical Coherence Tomography: Patients who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure will be approached for the study and enrolled if eligible.
  Optical Coherence Tomography: OCT will be performed with the St. Jude OCT system.
  Detection of metallic stent struts will be performed automatically with manual adjustments made as necessary. Stent area tracings will be automatically performed by interpolated contours connecting the center point of the luminal surface of each detected metallic strut. Stent expansion will be determined as the minimum stent area divided by the average reference lumen area and presented as a percentage. Neo-intimal hyperplasia (NIH) area will be determined in follow-up examinations as the area between the stent and lumen contours. Incomplete stent apposition (ISA) area will be determined as the area between the stent contour and the lumen contour at the site of malapposed struts, in a region not overlying a side branch ostium.
  Percent neointimal volume was mild with a median of 3.5% (IQR 2.3%-8.2%) at 3 months and 14.5% (IQR 13.5%-15.5%) at 12 months. The lumen was well preserved, and the median minimum lumen area (MLA) in the LM measured 9.97 mm2 (IQR 9.11 mm2 -10.37 mm2) at 3 months.
Arm/Group | Optical Coherence Tomography
Number analyzed (Participants) | 6
Participants | 4

4. Secondary Outcome: 12-month Persistent Stent Malapposition
Description: as for outcome 3
Time Frame: 12 month
Population: Participants with data analyzed at 12 months.
  1 out of 2 participants analyzed had malapposition at 12-month.
Measure: Count of Participants; unit: Participants
Groups:
- Optical Coherence Tomography: Patients who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure.
Arm/Group | Optical Coherence Tomography
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: MACE include:
  * Death
  * Myocardial infarction
  * Stroke (cerebrovascular accident or CVA)
  * Urgent revascularization
  * Repeat revascularization
  * Bleeding
  * Stent thrombosis
  * Rehospitalization
Time Frame: MACE reported at 12 months
Population: Participants with MACE reported at 12 months.
Measure: Count of Participants; unit: Participants
Groups:
- MACE: Participants who have undergone clinically-indicated PCI of LM where OCT was performed as part of the routine index procedure.
Arm/Group | MACE
Number analyzed (Participants) | 12
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 1, 3, 6 and 12 months.
Arm/Group | Optical Coherence Tomography
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optical Coherence Tomography (N=12)
Urinary Tract infection (Renal and urinary disorders) | 1 (1)
Stent mallaposition needing angioplasty (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optical Coherence Tomography (N=12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT03474432/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT03474432/ICF_001.pdf